CLINICAL TRIAL: NCT06334861
Title: Multidisciplinary Hospital-Territory Vaccine Center: a Model for Achieving the Herpes Zoster Vaccine Coverage
Acronym: CeVOT-Her-Zo
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5001
Record Dates: First submitted 2023-03-13; First posted 2024-03-28 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fragile patients vaccinated with herpes zoster vaccine: Patients with immunodeficiency and/or immunosuppression afferent to the U.O.C. Rheumatology, U.O.C. Hematology and Hematopoietic Stem Cell Transplantation, U.O.C. Infectious Diseases and Geriatric Internal Medicine, Travel Clinic and Occupational Health Outpatient Clinic of FPU Agostino Gemelli IRCCS who meet the inclusion criteria will be recruited.
  Inclusion Criteria.
  * Patients with congenital and/or acquired immunodepression;
  * Age > 18 years;
  * Signature of informed consent Exclusion criteria.
  * Persons younger than 18 years of age
  Interventions: Biological: Herpes Zoster adjuvanted recombinant vaccine

INTERVENTIONS:
Biological: Herpes Zoster adjuvanted recombinant vaccine — patients will receive two doses of vaccine with an interval between the first and second dose of 2 months

SUMMARY:
The National Vaccination Program, updated by the Ministry of Health in 2021, provides a new vaccination opportunity for frail patients against Herpes zoster virus (HZ). The new treatment option, on the other hand, is designed by combining VZV-specific antigen (gE) with an adjuvant system (AS01B) to induce antigen-specific cellular and humoral immune responses in individuals with preexisting immunity to VZV. Efficacy, assessed in people given two doses 2 months apart, is around 97% in those aged 50 years and 91% in those over 70 years. In the studies conducted, HZ-related hospitalizations were significantly reduced. The vaccine schedule calls for the administration of two doses 2 months apart. The current HZ Vaccination Program implemented at the regional level recommends its active and free offer in people from 18 years of age with congenital and/or acquired immunodepression, through a collaborative relationship involving, on the one hand, multispecialist and multiprofessional medical staff and, on the other hand, citizens called to play a role that is no longer passive but the subject of empowerment by consciously making their own health choices. The collaboration with ASL Roma1, in this sense, acquires value as guarantor of the supply of the adjuvanted recombinant anti-HZ vaccine and of the appropriate reporting of vaccination coverage, which to date is still far from the targets set by the PNPV'17-'19 in adults at risk for disease.

The purpose of this study Single-center prospective longitudinal observational cohort study is to verify patients' compliance with the proposed vaccination, the effectiveness of counseling carried out by a multidisciplinary team in the hospital setting.

DETAILED DESCRIPTION:
Vaccinations are a safe and effective means of protecting populations against specific infectious diseases and are recommended at all ages. The implementation of Vaccine Services also goes through the introduction of new modes of delivery, with pathways increasingly suitable to promote and implement the prevention campaign. The Hospital represents the place par excellence where categories of at-risk individuals are intercepted for whom adequate vaccine protection is a priority. A Hospital Vaccine Center (CVO), therefore, could effectively select patients/users in both a programmed and an opportunity and initiative medicine perspective, putting in place the national and regional indications that would like to integrate the vaccine offer with the clinical care pathways of at-risk categories that belong to different disciplines. In line with these provisions of the Ministry of Health and the Lazio Region, the CVO is also proposed as a referral structure for the immunization of patients with high clinical complexity in order to achieve optimization, personalization and compliance with the vaccine program of individuals at higher risk, who, due to underlying diseases or ongoing treatments, need monitoring of the antibody response and have an indication to be vaccinated in a protected environment.

In concert with a forward-looking vision of "Hospital as a Vaccine Care and Prevention Center," the optimal vaccination pathway should be built in collaboration with the territorial reality, becoming a strategic-cultural continuum of promoting vaccination both as individual protection of frail adults and as a solidaristic choice in the interest of the entire community. So, our project is proposed as an organizational synergy between the I.R.C.C.S. Policlinico Universitario A. Gemelli and ASL Roma 1 (relying on the agreement stipulated between ASL Roma 1 and Policlinico Gemelli Foundation, regarding the supply of vaccines), thus ensuring cultural confrontation between hygienists and specialists involved in the care of frailty, constituting a scientific training network of professionals dedicated to counseling and for the drafting of vaccine protocols dedicated to the various conditions of interest.

The Strategic Advisory Group of Experts (SAGE) of the World Health Organization (WHO) defines "vaccine hesitation" as a delay in acceptance or refusal of vaccination despite vaccine availability. In any case, it appears mandated to put in place all interventions aimed at raising awareness of the benefits of vaccination, counteracting misinformation, fears, and reticence. The strategic value of the "Hospital Vaccine Center" model-pilot is inherent in offering the best and most appropriate immunological prophylaxis, being able to seize the right time (with respect to clinical-diagnostic and therapeutic-surgical follow-ups), place and time most effective for both the user and the specialist, managing patient care, promoting technological and scientific innovativeness, collecting and generating data (immunogenicity, efficacy, safety, compliance) and integrated "vaccine therapy-prevention" operational protocols, all in a real-world setting in specific fragile populations. All this is done by leveraging the specialist-patient fiduciary relationship and facilitating the vaccine culture pathway that sees vaccine delivery integrated with patient care activities.

The purpose of this study Single-center prospective longitudinal observational cohort study is to verify patients' compliance with the proposed vaccination, the effectiveness of counseling carried out by a multidisciplinary team in the hospital setting.

Primary endpoint of the study is to verify patients' compliance to the vaccination proposal, in terms of the number of patients vaccinated compared to the total number of subjects eligible for vaccination and afferent to the participating OUs.

Secondary endpoint:

* To assess the vaccination coverage of subjects afferent to the FPU Agostino Gemelli IRCCS.
* Assess vaccination coverage (defined as the number of vaccinated patients compared to the total number of patients eligible for vaccination) stratified by the different diseases from which the subjects are affected.
* Assessment of adverse reactions in terms of number, type, and time of onset since administration of the first and second dose both overall and stratified by baseline disease, batch number of vaccine administered, and dose.
* Assessment of Vaccine Confidence in the hospital setting in terms of results extracted from validation of the VAX scale, both overall and stratified by the diseases they are affected by.
* Analysis of the economic impact of the anti-HZ vaccine pathway. Patients with immunodeficiency and/or immunosuppression afferent to the U.O.C. Rheumatology, U.O.C. Hematology and Hematopoietic Stem Cell Transplantation, U.O.C. Infectious Diseases and Geriatric Internal Medicine, Travel Clinic and Occupational Health Outpatient Clinic of the FPU Agostino Gemelli IRCCS who meet the inclusion criteria will be recruited.

Inclusion Criteria.

* Patients with congenital and/or acquired immunodepression;
* Age > 18 years;
* Signature of informed consent

The study involves 4 phases:

1. Implementation of an anti-HZ vaccine campaign from the date of approval of this study by the Local Ethics Committee at the Virtual CV afferent to the U.O.C. Hospital Hygiene of the Agostino Gemelli IRCCS University Polyclinic Foundation.
2. Vaccination slots will be sized according to requests from the Responsible Clinicians of individual DHs. Vaccinations will be administered in an ad hoc identified room in each individual DH one day/week from 8 am to 5 pm (4 vaccinations/h for a maximum of 40 vaccinations/day).
3. Treating physicians will be responsible for listing selected patients for vaccination on the dedicated day. The booster will be scheduled respecting the target eligible population deadline of 30 days between the first and second dose. The vaccinating physicians, assisted by a nurse, proceed with the collection of the pre-vaccination history and the administration of informed consent. Concurrently, the administration of the Vaccination Attitudes Examination Scale (VAX) questionnaire, an instrument validated in the literature for the study of "vaccine hesitancy," takes place. Then, the nurse administrators, with the supervision of the nursing coordinator, proceed with the administration of the vaccine. After administration, there is a waiting period of at least 15 minutes for surveillance of the occurrence of any adverse reactions for which appropriate medications and medical devices are provided.

   Suspected adverse reactions observed after vaccine administration will be reported to the Competent Authority AIFA, in accordance with the provisions of the current regulations DM April 30, 2015, according to the postmarketing pharmacovigilance flow (https://www.aifa.gov.it/content/segnalazioni-reazioni-avverse). Medical and nursing staff at the vaccine site will report suspected adverse reactions that occurred during the scheduled observation period or if they become aware of them. Vaccine recipients are required to report any adverse event, suspected adverse reaction, to the DH at which they received the vaccine and also to the treating physicians at the referring NICUs, either through their GP or spontaneously by arranging for the report to be sent to AIFA through the dedicated online platform (www.vigifarmaco.it) or other planned modality (https://www.aifa.gov.it/content/segnalazioni-reazioni-avverse).
4. Economic evaluation of the impact achieved by the vaccine campaign under study and data dissemination.

Simile sizing: Since this is a large-scale observational real-life study, and given the purely exploratory primary endpoint, formal sample sizing is not necessary. However, based on the data available from the referral departments for the past year, it is estimated to include, among the immunocompromised subjects covered by the recommendation to the anti-HZ vaccine campaign: 50 HIV+ patients, 50 onco-hematology subjects, 50 immunocompromised rheumatology subjects, 50 frail geriatric patients, and 50 patients from the Travel Clinic and Occupational Health Outpatient Clinic for a total of 250 patients. These numbers may be higher or lower depending on the supply of vaccine doses by ASL Roma 1.

statistic analysis: All variables under study will be assessed by descriptive statistical techniques. In detail, qualitative variables will be expressed as absolute frequencies and percentages. Quantitative variables, on the other hand, after checking their distribution using the Shapiro Wilk test, will be described as mean and standard deviation (SD) or median and interquartile range (IQR). Patients' compliance with the proposed vaccination will be expressed in terms of the number and percentage of patients vaccinated out of the total number of subjects eligible for vaccination and afferent to the participating OUs in the project. Potential associations between compliant and non-compliant subjects and the clinical and socio-demographic variables provided by the referring OUs will be assessed by means of the Chi-square test or Fisher's exact test for qualitative data. Quantitative data, on the other hand, will be assessed by Student's t test or Mann Withney's U test depending on the distribution of the data. Variables significantly associated with the univariable analysis will be included in a multivariable logistic regression model. The same analyses will be conducted, among the secondary endpoints, by stratifying the population into subgroups according to their disease classes. Adverse reactions to vaccines will be described in terms of absolute frequency and percentage of total doses administered and stratified by dose number (first or second). Their associations with underlying disease, concomitant drugs, time of onset from administration, batch number, and demographic variables will also be assessed using the statistical tests mentioned above. The economic impact related to the introduction of the Herpes-Zoster vaccine campaign will be evaluated through a budget impact analysis (BIA). Specifically, 2 alternative scenarios among them will be valued, and their results will be expressed in the form of differential resources associated with the scenarios under analysis. The perspective adopted is that of the institution (i.e., Fondazione Policlinico Universitario Agostino Gemelli IRCCS). Costs will be expressed in euros (€). The time horizon of the analysis will be medium to short (i.e., 1-5 years), in accordance with international guidelines. A cost-effectiveness evaluation will complement the BIA to simultaneously assess both costs and health outcomes associated with the presence of an anti-HZ vaccine pathway. In this case, both direct and indirect costs will be assessed. The perspective to be taken in this analysis will be that of society. Costs will be expressed in euros. All analyses will be conducted with R software version 4.1.2 (CRAN ®, R Core 2021).

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital and/or acquired immunodepression;
* Age > 18 years;
* Signature of informed consent

Exclusion Criteria:

* Persons younger than 18 years of age
* Pregnancy and lactation
* Hypersensitivity to the active ingredients and excipients in the formulation
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since this is a large-scale observational real-life study, and given the purely exploratory primary endpoint, formal sample sizing is not necessary. However, based on the data available from the referral departments for the past year, it is estimated to include, among the immunocompromised subjects covered by the recommendation to the anti-HZ vaccine campaign: 50 HIV+ patients, 50 onco-hematology subjects, 50 immunocompromised rheumatology subjects, 50 frail geriatric patients, and 50 patients from the Travel Clinic and Occupational Health Outpatient Clinic for a total of 250 patients. These numbers may be higher or lower depending on the supply of vaccine doses by ASL Roma 1.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Compliance to vaccination | 12 months
  Patients' compliance with the vaccination proposal, in terms of the number of patients vaccinated compared with the total number of subjects eligible for vaccination and afferent to the participating OUs in the project

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Laurenti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli - UCSC, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No